CLINICAL TRIAL: NCT03643471
Title: Role of Advanced Magnetic Resonance Imaging in Diagnosis of Idiopathic Temporal Lobe Epilepsy
Brief Title: Advanced Magnetic Resonance Imaging in Temporal Lobe Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa Anas Abou El-Kasem, Assistant lecturer, Assiut University
Other Study IDs: MRI in temporal lobe epilepsy
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Temporal Lobe Epilepsy
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Magnetic resonance imaging with advanced sequences including volumetry, spectroscopy and tractograpghy.

SUMMARY:
We aim to o evaluate the role of conventional and advanced MRI sequences in diagnosis of idiopathic temporal lobe epilepsy including identification and lateralization of epileptogenic focus.

DETAILED DESCRIPTION:
Patients with history of partial seizures with or without secondary generalization attending at outpatient clinic or admitted at Neurology department of Assuit University Hospital will be included in the study MRI study will be done for each patient. MR imaging will be performed on a 1.5-T MR imaging unit (Siemens, Sembra medical system,German).

Prospectively completed data forms will be analyzed and compared. Statistical tests appropriate to the nature of the data will be used.

All patients will not be subjected to risk of any kind during this study. All patients' data will be confidentially kept. Approval of the ethical committee of Faculty of Medicine, Assiut University.

An informed consent will be taken from all patients included in this study. The research will be conducted only by scientifically qualified and trained personnel.

The procedures included in this study have been already used in hospital and centers in and outside Egypt

ELIGIBILITY:
Inclusion Criteria:

* patients with history of partial seizures with or without secondary generalization attending at outpatient clinic or admitted at Neurology department of Assuit University Hospital will be included in the study based on the following criteria:

  * Clinical features consistent with seizures of temporal lobe origin.
  * Focal ictal temporal lobe patterns recorded with EEG.
  * No lesion detected by conventional MR imaging other than mesial temporal sclerosis.

Exclusion Criteria:

* Any general contraindication of MRI in some cases as presence of para magnetic substance as pacemakers or in patients with claustrophobia.
* Subjects with age less than 12 year old.
* Patients with any structural lesion other than mesial temporal sclerosis identified on MR brain imaging.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patients with history of partial seizures with or without secondary generalization attending at outpatient clinic or admitted at Neurology department of Assuit University Hospital with clinical features consistent with seizures of temporal lobe origin, Focal ictal temporal lobe patterns recorded with EEG and no lesion detected by conventional MR imaging other than mesial temporal sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Calculating the sensitivity,specificity and accuracy of hippocampal volumetry , T2 relaxometry , MR spectroscopy and diffusion tensor imaging in identification and lataeralization of epileptogenic focus | baseline
  * Quantification of hippocampal volumes bilaterally by mean of hippocampal volumetry
  * Change in metabolites ratio at the affected hippocampus by mean of MR spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Muhlhofer W, Tan YL, Mueller SG, Knowlton R. MRI-negative temporal lobe epilepsy-What do we know? Epilepsia. 2017 May;58(5):727-742. doi: 10.1111/epi.13699. Epub 2017 Mar 7. PMID 28266710
- [Background] Crocker CE, Pohlmann-Eden B, Schmidt MH. Role of neuroimaging in first seizure diagnosis. Seizure. 2017 Jul;49:74-78. doi: 10.1016/j.seizure.2016.05.015. Epub 2016 Jun 1. PMID 27324840
- [Background] Ruber T, David B, Elger CE. MRI in epilepsy: clinical standard and evolution. Curr Opin Neurol. 2018 Apr;31(2):223-231. doi: 10.1097/WCO.0000000000000539. PMID 29389747
- [Background] Chinchure S, Kesavadas C, Thomas B. Structural and functional neuroimaging in intractable epilepsy. Neurol India. 2010 May-Jun;58(3):361-70. doi: 10.4103/0028-3886.65569. PMID 20644262